CLINICAL TRIAL: NCT02552199
Title: A Non-Interventional Study To Assess Sweating, As Measured By Gravimetry, In Subjects With Primary Hyperhidrosis And In Healthy Individuals
Brief Title: A Non-Interventional Study To Assess Sweating
Status: Completed | Type: Observational
Sponsor: Botanix Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: BBI-4000-EM-101
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Results first posted 2023-10-23 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- with hyperhidrosis: Patients with primary palmar hyperhidrosis
  Interventions: Other: gravimetric
- healthy: Healthy adult patients
  Interventions: Other: gravimetric

INTERVENTIONS:
Other: gravimetric

SUMMARY:
To evaluate the gravimetric sweat measurements in subjects who meet the subjective criteria for a diagnosis of palmar hyperhidrosis compared to subjects without hyperhidrosis.

DETAILED DESCRIPTION:
This is a Non-Interventional Study To Assess Sweating, As Measured By Gravimetry, In Subjects With Primary Hyperhidrosis And In Healthy Individuals .

The objective of this study is to determine the threshold gravimetric measurement for subjects with palmar hyperhidrosis.

ELIGIBILITY:
Inclusion Criteria:

* Females should not be pregnant or lactating.
* For subjects with palmar hyperhidrosis: Primary palmar hyperhidrosis of at least 6 months's duration and Hyperhidrosis disease severity score of 3 or 4 at baseline
* For healthy participants: no history or current report of hyperhidrosis and Hyperhidrosis disease severity score of 1 at baseline

Exclusion Criteria:

* Recent therapeutic interventions or treatments for palmar hyperhidrosis
* Any major illness within 30 days before the screening
* Females who are pregnant, lactating, or planning a pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with palmar hyperhidrosis and healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia S Walker, M.D.,Ph.D., Study Director — Botanix Pharmaceuticals
Locations (1):
- Carpinteria Dermatology, Carpinteria, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- With Hyperhidrosis: Patients with primary palmar hyperhidrosis
  gravimetric
- Healthy: Healthy adult patients
  gravimetric
Period: Overall Study
Arm/Group | With Hyperhidrosis | Healthy
Started | 17 | 11
Completed | 17 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | With Hyperhidrosis | Healthy | Total
Number analyzed (Participants) | 17 | 11 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.59 (16.33) | 47.91 (14.50) | 43.46 (15.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 20
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 12 | 7 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 10 | 19
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Mean Average (Standard Deviation) Total Palmar Gravimetric Sweat Production (GMSP) Between Subject Groups (Adult Patients With Hyperhidrosis Versus Healthy Adult Volunteers).
Description: Gravimetric assessments were conducted in a temperature controlled room on two separate occasions over a five minute period (two assessments/palm), assessing both palms. An individual palm GMSP was determined by subtracting the Weight (g) of individual gauze in contact with palm after five minutes - Weight (g) of individual gauze prior to palmar contact. For this analysis, each participant could provide two results (1 Total GMSP/occasion) as:
  Total GMSP 1 [g] = Right palm GMSP 1 [g] + Left palm GMSP 1 [g] Total GMSP 2 [g] = Right palm GMSP 2 [g] + Left Palm GMSP 2 [g] Mean average [g] (standard deviation) Total GMSPs were compared between Subject Groups (adult patients with hyperhidrosis versus healthy adult volunteers).
Time Frame: Gravimetric assessments were conducted in a temperature controlled room on two separate occasions over a five minute period (two assessments/palm), assessing both palms.
Population: Full analysis set including all enrolled subjects.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | With Hyperhidrosis | Healthy
Number analyzed (Participants) | 17 | 11
grams | 0.7687 (0.8300) | 0.1762 (0.1010)

ADVERSE EVENTS:
Time Frame: 14 days
Description: Due to the short duration and non-interventional nature of the study, only procedure-related AEs were collected.
Arm/Group | With Hyperhidrosis | Healthy
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/11
Other Adverse Events (participants affected / at risk) | 0/17 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes